CLINICAL TRIAL: NCT05440799
Title: Safety, Tolerability and Pharmacokinetics of Multiple Rising Oral Doses of BI 1819479 in Healthy Female Subjects of Non-childbearing Potential (Double-blind, Randomised, Placebo-controlled, Parallel Group Design)
Brief Title: A Study to Test How Healthy Women Tolerate Different Doses of BI 1819479
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1462-0002; 2021-006992-41 (EudraCT Number)
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BI 1819479 (Experimental)
  Interventions: Drug: BI 1819479
- Placebo (Placebo Comparator)
  Interventions: Drug: BI matching placebo

INTERVENTIONS:
Drug: BI 1819479 — BI 1819479
  Arms: BI 1819479
Drug: BI matching placebo — BI matching placebo
  Arms: Placebo

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 1819479 in healthy female subjects of non-childbearing potential.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non-childbearing potential according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age between 18 years and 67 (inclusive)
* Body mass index (BMI) of 18.5 to 30.9 (weight divided by height squared)(kg/m2) (inclusive)
* Signed and dated written informed consent in accordance with International Conference on Harmonisation (ICH) - Good Clinical Practice (GCP) and local legislation prior to admission to the trial
* Female subject of non-childbearing potential defined as:

  * Permanently surgically sterilised (hysterectomy, bilateral salpingectomy and/or bilateral oophorectomy)
  * Postmenopausal, defined as no menses for 1 year in women aged = 51 years or no menses for 2 years in women aged = 50 years, without an alternative medical cause
  * In questionable cases of postmenopausal status:

    * Women not using sex hormone medication such as hormone replacement therapy may be included if a blood sample confirms levels of Follicle-stimulating hormone (FSH) > 40 unit/liter (U/L) and estradiol < 30 nanogram per liter (ng/L)
    * Women using sex hormone medication such as hormone replacement therapy cannot be included in the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimetres of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Further exclusion criteria apply

Ages: 18 Years to 67 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2023-08-02 (Actual)

PRIMARY OUTCOMES:
Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator | up to 106 days

SECONDARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) | up to 92 days
Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmax,ss) | up to 92 days

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https:// www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com